CLINICAL TRIAL: NCT06113302
Title: A Pilot, Open-Label Study of Luspatercept for Patients With Lower Risk Myelodysplastic Syndromes (MDS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-1080; NCI-2023-09312 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants with lower risk MDS patients who have symptomatic anemia that are transfusion independent (TI). Participants will be asked to come to the study clinic weekly for the first 3 weeks and then 1 time every 3 weeks after that to have tests and procedures (such as physical exams and blood draws). Luspatercept will be administered once every 3 weeks.
  Interventions: Drug: Luspatercept
- Cohort 2 (Experimental): Participants with lower risk MDS that are transfusion dependent (TD). Participants will be asked to come to the study clinic weekly for the first 3 weeks and then 1 time every 3 weeks after that to have tests and procedures (such as physical exams and blood draws). Luspatercept will be administered once every 3 weeks.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Given by SC or (Injection)
  Other Names: ACE-536

SUMMARY:
To learn if luspatercept is more effective in helping to reduce the number of blood transfusions needed by patients with LR-MDS.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives:

* To assess the clinical activity and safety of luspatercept in patients with transfusion independent lower risk MDS
* To assess the clinical activity and safety of luspatercept in patients with transfusion dependent lower risk MDS
* To study the effects on hematopoeisis of luspatercept in patients treated on this study

Secondary Objectives:

* To assess the duration of response of patients with treated with luspatercept in this study
* To assess the overall survival and time to transformation of patients with treated with luspatercept in this study
* To assess transfusion free survival period in patients that were transfusion independent treated with luspatercept in this study
* To measure trends in neutrophil and platelet counts in patients treated in this study

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; as MDS there is no significant experience with luspatercept in pediatric patients
2. Cohorts #1 and #2: Diagnosis of MDS according to WHO 2023 criteria (5) and with low or int-1 risk by IPSS or a score of ≤ 3.5 by IPSS-R.(3, 22)
3. Cohort #2: Patient defined as transfusion dependent by documentation of receiving at least 2 units of packed red blood cells (PRBCs) for a hemoglobin of less than 8.0 g/dL during an 8-week period prior to study enrollment.
4. Cohort #1: Patients with symptomatic anemia that are transfusion independent defined as not requiring a transfusion for a hemoglobin of less than 8.0 g/dL during an 8-week period prior to study enrollment.
5. MDS patients with either a platelet count of ≤100 K/uL and/or ANC of ≤1.8 K/uL
6. Patient must have signed an informed consent and is willing to participate in the study.
7. Adequate hepatic function with total bilirubin ≤3 x ULN, AST or ALT ≤3xULN.
8. Serum creatinine clearance ≥40mL/min and no end/stage renal disease (using Cockcroft-Gault).
9. ECOG performance status </=2.

Exclusion Criteria:

1. Active infection not adequately responding to appropriate antibiotics.
2. Prior treatment with luspatercept or sotarcetept
3. Female patients who are pregnant or lactating.
4. Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study. Reproductive potential is defined as no previous surgical sterilization or females that are not post-menopausal for 12 months.
5. Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening.
6. History of an active malignancy within the past 2 years prior to study entry, with the exception of: a. Adequately treated in situ carcinoma of the cervix uteri b. Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin or any other malignancy with a life expectancy of more than 2 years.
7. Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy (within 14 days of initiating study treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org